CLINICAL TRIAL: NCT05377333
Title: Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3457263 Alone and in Combination With GLP-1 RA in Patients With Type 2 Diabetes
Brief Title: A Study of LY3457263 Alone and in Combination With Dulaglutide (LY2189265) in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18129; J1R-MC-GZFB (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-05-16; First posted 2022-05-17 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3457263 (Alone) (Experimental): LY3457263 administered subcutaneously (SC).
  Interventions: Drug: LY3457263
- Placebo (Alone) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo
- LY3457263 + Dulaglutide (Experimental): LY3457263 in combination with dulaglutide administered SC.
  Interventions: Drug: LY3457263; Drug: Dulaglutide
- Placebo + Dulaglutide (Experimental): Placebo in combination with dulaglutide administered SC.
  Interventions: Drug: Placebo; Drug: Dulaglutide

INTERVENTIONS:
Drug: LY3457263 — Administered SC.
  Arms: LY3457263 (Alone); LY3457263 + Dulaglutide
Drug: Placebo — Administered SC.
  Arms: Placebo (Alone); Placebo + Dulaglutide
Drug: Dulaglutide — Administered SC.
  Other Names: LY2189265
  Arms: LY3457263 + Dulaglutide; Placebo + Dulaglutide

SUMMARY:
The main purpose of this study is to investigate the safety and tolerability of the study drug LY3457263 when administered alone or in combination with glucagon-like peptide 1 (GLP-1) receptor agonist (RA) in participants with type 2 diabetes. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. The study will last up to approximately 16 weeks excluding the screening period for each participant and include up to 17 visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants with type 2 diabetes (T2D) at least 6 months before screening
* Participants treated for T2D with diet and exercise, with or without metformin
* Have a glycated hemoglobin A1c (HbA1c) value of ≥ 7.5% and ≤10.5%
* Have had a stable body weight for 3 months and body mass index (BMI) of 27.0 to 45.0 kilograms per meter squared (kg/m²)
* Male participants who agree to use effective methods of contraception and female participants not of childbearing potential

Exclusion Criteria:

* Have a history of or current cardiovascular, respiratory, hepatic, renal, GI, endocrine (apart from T2D), hematological, or neurological disorders capable of altering the absorption, metabolism, or elimination of drugs
* Have type 1 diabetes mellitus or latent autoimmune diabetes in adults or maturity-onset diabetes of the young
* Have a history of proliferative diabetic retinopathy, diabetic maculopathy, or severe non-proliferative diabetic retinopathy
* Have known allergies to GLP-1 receptor agonists

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Predose up to 16 weeks
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3457263 | Pre-dose on Day 1 up to 85 days post-dose
  PK: AUC of LY3457263

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - CenExel ACT, Anaheim, California
  - Qps-Mra, Llc, South Miami, Florida
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - CenExel-HRI, Berlin, New Jersey

IPD SHARING:
Plan to Share IPD: No